CLINICAL TRIAL: NCT03020784
Title: A Phase 1, Randomized, Double-blind, Sponsor-open, Placebo-controlled, Single-ascending Dose Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of Pf-06818883 Following Single Intravenous Administration In Healthy Subjects
Brief Title: Safety and Tolerability of PF-06818883 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated on 16JUN2017 for safety reasons
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: C0601001
Record Dates: First submitted 2016-10-27; First posted 2017-01-13 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: acute neuroinflammatory

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): IV placebo
  Interventions: Drug: Placebo
- PF-06818883 (Experimental): Experimental drug
  Interventions: Drug: PF-06818883

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: PF-06818883 — Treatment
  Arms: PF-06818883

SUMMARY:
Safety, Tolerability and Pharmacokinetics of PF-06818883

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of nonchildbearing potential and/or male subjects
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Any condition possibly affecting the placement of an intravenous drug administration line.
* A confirmed positive urine drug screen
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day or 2 chews of tobacco per day
* Treatment with an investigational drug within 30 days (or as determined by the local requirement)
* Screening supine blood pressure >140 mm Hg (systolic) or <90 mm Hg (diastolic), following at least 5 minutes of supine rest
* Screening supine 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* History of human immunodeficiency virus (HIV), hepatitis B or C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb) or hepatitis C antibody (HCVAb).
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Change in Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 0, Day 1, Day 2, Day 3
  An assessment of Adverse Events
Change in Physical examination | Day 0, Day 1, Day 2 and Day 3
  Safety test to check overall health
Change in Neurological Exam | Day 0, Day 1, Day 2 and Day 3
  Assessment of sensory neuron and motor responses
Change in 12-lead ECG (electrocardiogram) | Day 1 hr 0.25, 1, 2, 6, 8, 12, Day 2 hr 24 and 36, Day 3 hr 48
  heart's electrical activity recorded from electrodes on the body surface
Change in Vital signs | Day 1 hr 0.25, 1, 2, 6, 8, 12, Day 2 hr 24 and 36, Day 3 hr 48
  clinical measurements, specifically pulse rate, temperature, and blood pressure, that indicate the state of a patient's essential body functions
Change in Clinical laboratory tests (haematology: haemoglobin; haematocrit/erythrocytes; haemoglobin/erythroctes; Erythro-, leuco-,lympho-, mono-Cytes; Platelets) | Day 0, Day 2 and Day 3
  Intended to detect, identify, or quantify one or more significant substances, evaluate organ functions, or establish the nature of a condition

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) after single dose for all periods | Day 1 hr 0.25, 0.5, 1, 1.5, 2, 3, 6, 8, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48
  Cmax after a single dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) after single dose for all periods | Day 1 hr 0.25, 0.5, 1, 1.5, 2, 3, 6, 8, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48
  Tmax after single dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) after single dose for all periods | Day 1 hr 0.25, 0.5, 1, 1.5, 2, 3, 6, 8, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) after single dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] after single dose for all periods | Day 1 hr 0.25, 0.5, 1, 1.5, 2, 3, 6, 8, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48
  AUC (0 - inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf) after single dose
Plasma Decay Half-Life (t1/2) after single dose for all periods | Day 1 hr 0.25, 0.5, 1, 1.5, 2, 3, 6, 8, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half after single dose
Clearance (CL) after single dose for all periods | Day 1 hr 0.25, 0.5, 1, 1.5, 2, 3, 6, 8, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Volume of Distribution (Vss) after single dose for all periods | Day 1 hr 0.25, 0.5, 1, 1.5, 2, 3, 6, 8, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48
  Volume of distribution is defined as the volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Dose-Normalized Maximum Plasma Concentration (Cmax(dn)) after single dose for all period | Day 1 hr, 0.25, 0.5, 1, 1.5, 2, 3, 6, 8, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48
  Dose-Normalized Cmax after a single dose
Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast(dn)) after single dose for all periods | Day 1 hr 0.25, 0.5, 1, 1.5, 2, 3, 6, 8, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48
  Dose Normalized Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast(dn)) after single dose
Dose Normalized Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf(dn))] after single dose for all periods | Day 1 hr 0.25, 0.5, 1, 1.5, 2, 3, 6, 8, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48
  AUC (0 - inf (dn)) = Dose Normalized Area under the plasma concentration versus time curve (AUC(dn)) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf) after single dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C0601001&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Sponsor-open%2C+Placebo-controlled%2C+Single-ascending+Dose+Study+To+Evaluate+The+Safety%2C+Tolerability+And+Pharmacokinetics+Of+Pf-06818883+Following+Single+Intravenous+Administration+In+Healthy+Subjects